CLINICAL TRIAL: NCT02157987
Title: Treatment of Hereditary Hemorrhagic Telangiectasia of the Nasal Mucosa by Intranasal Bevacizumab : Search for Effective Dose
Acronym: EROSB
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2013-004390-27
Record Dates: First submitted 2014-06-04; First posted 2014-06-06 (Estimated); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Telangiectasia, Hereditary Hemorrhagic
Keywords: telangietasia hereditary hemorragic; epistaxis; safety; quality of life; bevacizumab; spray
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic; Epistaxis

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- bevacizumab (Experimental): bevacizumab spray
  Interventions: Drug: bevacuzimab spray

INTERVENTIONS:
Drug: bevacuzimab spray

SUMMARY:
Epistaxis are present in over 90 % of patients with Rendu - Osler . They involve no significant difference 2 sexes. They often appear in childhood and adolescence and are present in three-quarters of patients at the age of 20 years. These epistaxis increasing in frequency and volume to the age of 60 in 2/3 of patients. Epistaxis are spontaneous , repetitive and recurring . They are highly variable in duration, intensity and frequency of occurrence . Some patients may have more than 40 monthly episodes with mean duration of 5 minutes of bleeding and chronic anemia and can sometimes acute anemia with transfusions need to be source. These epistaxis stigmatize patients and inevitably affect their quality of life and social skills . The various proposed ( cauterization , intra- mucosal injections, laser selective hémostatses , embolization or surgical dermoplasties ) allow for some short-term remissions . Bevacizumab is an antiangiogenic use in the treatment of colorectal cancers . It is also used in ophthalmology intravitreal to reduce vascular proliferation in glaucoma retinopathy and certain corneal neovascularization. In 2009, Prithviraj reported the use of bevacizumab injection to treat pulmonary arteriovenous malformations in a patient with Rendu - Osler . The result is doubly interesting including a saving action on epistaxis which decrease in frequency and duration. This communication prompted the authors to focus more on this medication. The product has been used in local submucosal injection intranasal laser was coupled with satisfactory results objectified by a decrease in the number of epistaxis , reducing blood transfusions and improved social lives. The use of local instillation bevacuzimab represents a way forward for the treatment of these epistaxis.

ELIGIBILITY:
Inclusion Criteria:

* patients with Rendu-Osler-Weber disease
* patients with iterative epistaxis (at least 10 per month)
* patients without treatment for 3 months with usual techniques (for the epistaxis)
* patients speaking french fluently
* patients with written consents
* affiliation to social security
* women with effective contraception during the treatment and for 6 months after stopping

Exclusion Criteria:

General criteria:

* Pregnant women, breastfeeding
* Hypersensitivity to the active substance or any of its excipients
* Hypersensitivity to the products of Chinese hamster ovary cells or other human or humanized recombinant antibodies
* Inability to undergo medical monitoring due to reasons geographical, social or psychological
* Patient under guardianship
* Patient included in another biomedical research protocol

Related to medical history criteria:

* Uncontrolled hypertension ( systolic BP > or = 150 mmHg and / or Diastolic BP > or = 100 mmHg)
* Thrombocytopenia <100 G / L
* Taking NSAIDs within ten days prior to inclusion
* Anticoagulant therapy or thrombolytic within 28 days before inclusion
* Tumor, genetic predisposition to bleeding, coagulopathy , patient receiving treatment full anticoagulant dose for an event thromboembolism prior to inclusion
* Major surgery within 28 days prior to inclusion
* History of thromboembolic disease within 6 months prior to enrollment
* Arteriovenous malformation localized to the brain, liver or lung on scanner older than 5 years
* History of heart failure
* Patients with proteinuria / creatinine greater than 2g / g

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-12-15 (Actual); Primary Completion 2020-10-08 (Actual); Study Completion 2021-12-08 (Actual)

PRIMARY OUTCOMES:
decrease of at least 50% of number of epistaxis in a month compared to the month before inclusion. | one month

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Caen, Caen, France